CLINICAL TRIAL: NCT06078878
Title: Clinical Feasibility Evaluation of the Gentuity HF-OCT Imaging System With Vis-M Micro-Imaging Catheter
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gentuity, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 003818
Record Dates: First submitted 2023-10-02; First posted 2023-10-12 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Anatomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Neurovascular Imaging (Experimental): Use of the Gentuity HF-OCT Imaging System with Vis-M Micro-Imaging Catheter ("Gentuity Neurovascular Imaging System") as a diagnostic tool for intravascular imaging in the cerebrovasculature.
  Interventions: Device: HF-OCT Imaging System with Vis-M Micro-Imaging Catheter

INTERVENTIONS:
Device: HF-OCT Imaging System with Vis-M Micro-Imaging Catheter — Subjects undergo HF-OCT imaging of the desired intravascular segement

SUMMARY:
This study is a prospective, single arm, unblinded, and open-label study. The study is designed to evaluate the use of the Gentuity Neurovascular Imaging System in patients undergoing elective neurointerventional diagnostic procedures.

DETAILED DESCRIPTION:
Patients undergoing elective, neurointerventional procedures, or patient undergoing follow-up diagnostic procedures who meet all inclusion criteria and none of the exclusion criteria will be considered for enrollment. The study investigates the use of the Gentuity Neurovascular Imaging System as a diagnostic tool for intravascular imaging in the cerebrovasculature. The study evaluates the incidence and severity of device-related adverse events, clinical usability performance and technical performance of imaging quality.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are electively scheduled for either a follow-up cerebral angiogram or a diagnostic angiogram and may be candidates for a neuroendovascular procedure
* Patients that present with a Modified Rankin Score (mRS) ≤3
* Patients 18 years of age or older
* Patients willing and able to provide written informed consent to participate in evaluation

Exclusion Criteria:

* Patients with serious concurrent medical conditions including bacteremia or sepsis, acute renal failure at the time of the procedure, and major coagulation system abnormalities that in the opinion of the investigator could significantly increase risk
* Pregnant
* Patient has a known hypersensitivity to contrast media
* Patients undergoing an urgent or emergent neurointerventional procedure
* Patients that present with a Modified Rankin Score (mRS) ≥4
* Patients that present with an unresolved spontaneous subarachnoid hemorrhage and/or intracranial hemorrhage
* Participation in another clinical trial of an investigational drug or device
* Patient has existing Flow Re-Direction Endoluminal Device (FRED®) System

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Device Safety | 7 days
  Incidence and severity of device-related adverse events.

SECONDARY OUTCOMES:
Clinical performance | 1 day
  Operator evaluation of performance via Likert scale.
Technical performance | 1 day
  Clear image length (CIL) of the vessel

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Lylyk, MD, Principal Investigator — Clínica La Sagrada Familia
Locations (1):
- Clínica La Sagrada Familia, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No